CLINICAL TRIAL: NCT05518578
Title: RENAISSANCE Study: A Phase 2, Multicenter, Open Label Safety and Tolerability Study of SPN-817 in Adult Patients With Treatment Resistant Epilepsy
Brief Title: Safety and Tolerability Study of SPN-817 in Adult Patients With Treatment Resistant Epilepsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 817P202
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy; Seizures, Epileptic
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-Label Treatment (Experimental): 0.25 mg to 4 mg SPN-817 taken orally twice daily
  Interventions: Drug: SPN-817

INTERVENTIONS:
Drug: SPN-817 — oral capsule
  Other Names: (-)-Huperzine A extended-release

SUMMARY:
This study will evaluate the safety and tolerability of SPN-817 in adults with treatment resistant seizures

DETAILED DESCRIPTION:
This is a multicenter, three-phase, long-term open-label study assessing the safety and tolerability of SPN-817 in adults 18-70 years of age with treatment resistant epilepsy. The Screening period is up to 8 weeks in duration. For eligible participants, Treatment period is 20 weeks in duration followed by an optional Open-Label Extension period which is up to 52 weeks in duration.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of treatment resistant epilepsy as adjudicated by the Epilepsy Study Consortium.
2. Is male or female, aged 18 to ≤ 70 years at screening.
3. Is able to read, understand, and sign the Informed Consent Form (ICF). If the participant is unable to sign informed consent, a Legally Authorized Representative (LAR) will complete the ICF.
4. Ability to keep accurate seizure diaries (with the aid of a caregiver as needed).
5. Weight within the normal or overweight ranges according to accepted values of the Body Mass Index Chart (18.0 to 35 kg/m2).
6. Is able to swallow capsules whole without crushing, chewing, or cutting.
7. Is willing to adhere to all study procedures and able to attend study visits within the specified time windows.
8. Failure of at least 2 tolerated, appropriately chosen and adequately dosed ASM drug schedules to achieve sustained seizure freedom.
9. Taking at least 1 ASM at Screening and Baseline.
10. At least 4 seizures accepted by the Epilepsy Study Consortium for the secondary outcome (adjudicated as "probable seizures" that are countable) during the 42-day baseline seizure diary period, and no more than a 21-day period that was seizure-free.
11. A clinical diagnosis of Focal Cortical Dysplasia (FCD) Type I or Type II (approximately n=10) confirmed by:

    1. Likely FCD supported by neuroimaging that has been performed in the last 5 years, or
    2. History of surgical resection of the cortical dysplasia that is histopathologically confirmed in patients who continue to have uncontrolled seizures without a compelling alternate explanation for ongoing seizures.

    Note: The Epilepsy Study Consortium will review to confirm FCD/probable FCD diagnosis.
12. Be in good general health in the judgment of the PI based upon medical history, physical examination, standard 12-lead ECG, and clinical laboratory evaluations obtained during the Screening Period
13. Be able to comply with all study-specified procedures.
14. Non-pregnant females of childbearing potential (FOCP) who are either sexually inactive (abstinent) or, if sexually active with a male partner who is biologically capable of having children, must agree to use one of the following acceptable birth control methods beginning 30 days prior to the first dose of SPN-817, throughout the study, and for 30 days following the last dose:

    1. Simultaneous use of male condom and intra-uterine contraceptive device (IUD) placed at least 4 weeks prior to first SPN-817 administration
    2. Surgically sterile male partner
    3. Simultaneous use of male condom and diaphragm with spermicide
    4. Established hormonal contraceptive

    Females are considered not to be of childbearing potential if they are either post-menopausal (amenorrhea for at least 2 years and serum follicle stimulating hormone [FSH] level of >40 IU/L) or permanently sterilized (e.g., bilateral tubal ligation, hysterectomy, bilateral oophorectomy) for 6 months minimum.
15. Males must:

    1. Use 2 methods of contraception in combination if his female partner is of childbearing potential; this combination of contraceptive methods must be used from the Screening Visit to ≥ 1 month after the last dose of SPN-817, or
    2. Have been surgically sterilized prior to the Screening Visit.
    3. Refrain from donating any sperm until completion of the EOS Visit.
16. Patients who were previously enrolled in the BNI-02-1b FIAS study and benefited from the treatment, following the approval by both the PI and the sponsor to be enrolled in this study.

Exclusion Criteria:

1. Has taken huperzine A within the past year, with the exception of patients who were previously enrolled in the BNI-02-1b FIAS study, benefited from the treatment, and approved by the PI and the sponsor to be enrolled in this study.
2. Is planning to become pregnant or impregnate spouse, not using an acceptable method of birth control (defined as use of double-barrier birth control methods, use of oral contraceptives, or surgical sterilization), pregnant, or nursing.
3. Patients with combined focal and generalized syndrome as evidenced by severe developmental delay and multiple seizure types, confirmed by EEG (e.g., Lennox-Gastaut syndrome). Patient should also be excluded in case of non-diagnostic information.
4. Has non-epileptic events that could be confused by the patient and/or study staff as epileptic seizures.
5. Has only seizures that are difficult to count; for example, has seizures that are not clinically observable.
6. Has a history of only seizure clusters, for example, seizure clusters defined as multiple seizures with at least one seizure within 30 minutes of the previous seizure.
7. Has a history of status epilepticus in the 6 months prior to Screening.
8. Change in ASM regimen in the last 28 days prior to Screening. No changes in ASMs are allowed throughout the study period.
9. Vagus nerve stimulation (VNS), deep brain stimulation (DBS), responsive neurostimulator system (RNS), or other neurostimulation for epilepsy device implanted or activated <1 year prior to Screening; stimulation parameters that have been stable for <3 months; battery life of unit not anticipated to extend for duration of trial; or epilepsy surgery <1 year prior to Screening.
10. Active suicidal plan/intent in the past 6 months, or a history of suicide attempt in the last 2 years, or more than 1 lifetime suicide attempt. History of suicidal ideation.
11. Any condition that may impact a patient's ability to follow study procedures or a patient's safety, based on what is known about the pharmacology/toxicology profile of the trial agent(s).
12. Has a pre-existing medical condition (including an existing progressive or degenerative neurological disorder including brain tumor, active encephalitis, active meningitis or abscess) or takes medications that, in the PI's opinion, could interfere with the patient's suitability for participation in the study.
13. Has a history or evidence of current significant psychiatric disturbance (e.g., schizophrenia, schizoaffective, or bipolar disorder) that would preclude meaningful participation in the study procedures.
14. A history in the past 2 years or evidence of current alcohol and/or substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders 5th edition.
15. Has had any clinical laboratory abnormalities within the 2 months prior to screening considered of clinical significance by the PI.
16. Is HIV/Hepatitis B/Hepatitis C positive or has a positive urine drug screen.
17. Tobacco use as indicated by >5 cigarettes per week or the equivalent, 30 days prior to Day -1.
18. Is on concomitant therapy with non-ASMs that are cholinergic.
19. Is currently taking or within the 3 days prior to enrollment has taken Epigallocatechin gallate (EGCG); or consumed foods or drinks containing EGCG, including green, white, or oolong teas and certain black teas, or food containing >100 grams of carob powder. EGCG cannot be consumed throughout the study.
20. Has participated in any clinical investigational drug or device study within 4 weeks prior to study entry or within 5 half-lives of the clinical investigational drug, whichever is longer.
21. Clinically significant cardiologic abnormalities at Screening. One repeat assessment is allowed per investigator discretion.

    1. Abnormal ECG that is, in the investigator's opinion, clinically significant including heart rate (HR) <50 bpm (average of 3 recordings)
    2. PR interval > 220 ms
    3. QRS interval ≥ 120 ms
    4. QTcF (QT corrected for heart rate using Fridericia's method) interval > 450 ms for males and interval > 475 ms for females
    5. Second or third-degree atrioventricular block
    6. Any rhythm, other than sinus rhythm, that is interpreted by the investigator to be clinically significant
22. Creatinine clearance < 90 mL/min, according to the Cockcroft-Gault equation at Screening.
23. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or HR less than 50 or over 100 bpm) at Screening.
24. Patient has had greater than 2 allergic reactions to an ASM or one serious hypersensitivity reaction to an ASM.
25. Patients who donated 50 to 499 mL of blood within 30 days or more than 499 mL within 56 days prior to Day 1 dosing or have hemoglobin <128 g/L (males) or <115 g/L (females) and hematocrit <0.37 L/L (males) or <0.32 L/L (females) at Screening. Following screening and throughout the study, patient should not donate blood.
26. Any reason which, in the opinion of the PI, would prevent the patient from participating in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Effects of SPN-817 on safety and tolerability | 72 weeks
  The incidence of adverse events.

SECONDARY OUTCOMES:
Effect of SPN-817 on the motor seizure frequency | 72 weeks
  Percent change from baseline in quantifiable motor seizure frequency per 28 days during treatment in the combined Titration/Optimization and Maintenance Periods, in the Maintenance Period, and in the combined Maintenance and Open-Label Extension Periods. A "quantifiable motor seizure" is defined as a seizure adjudicated as probable and countable by the Epilepsy Study Consortium, Inc. (ESCI).
Effect of SPN-817 on the motor seizure frequency treatment response rate | 20 weeks
  The 30%, 50% and 75% motor seizure frequency treatment response rate during treatment in the combined Titration/Optimization and Maintenance Periods and in the Maintenance Period. The 30%, 50% or 75% seizure frequency treatment response rate is defined as the percent of subjects who have a ≥30%, ≥50%, or ≥75% reduction, respectively, in the change from baseline quantifiable motor seizure frequency. A "quantifiable motor seizure" is defined as a seizure adjudicated as probable and countable by the Epilepsy Study Consortium, Inc. (ESCI).
Effect of SPN-817 on seizure-free rate | 20 weeks
  The seizure free rate observed during treatment in the Maintenance Period and in the combined Titration/Optimization and Maintenance Periods. Seizure free rate is defined as the percent of subjects who do not experience a seizure during the designated period or the period of time.
Effect of SPN-817 on time to event analysis | 64 weeks
  The duration of time (days) elapsed between the start of the clinically relevant dose (maintenance period) and the time that the patient returns to baseline seizure frequency.
Effect of SPN-817 on incidence of motor seizure-free days. | 72 weeks
  Change from Baseline in the percentage of quantifiable motor seizure-free days per 28 days during treatment. A "quantifiable motor seizure" is defined as a seizure adjudicated as probable and countable by the Epilepsy Study Consortium, Inc. (ESCI).
Effect of SPN-817 on the Clinical Global Impression - Improvement (CGI-I) scale | 72 weeks
  CGI-I score by visit during treatment.
Effect of SPN-817 on the Clinical Global Impression - Severity (CGI-S) scale | 72 weeks
  Change from Baseline in the CGI-S score by visit during treatment.
Effect of SPN-817 on the Quality of Life in Epilepsy (QOLIE-31-P; v2.0) questionnaire | 72 weeks
  Change from Baseline in QOLIE-31-P score by visit during treatment.
Effect of SPN-817 on the Seizure Related Disability Assessment Scale (SERDAS) scale | 72 weeks
  Change from Baseline in SERDAS score by visit during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, MBA, Study Director — Supernus Pharmaceuticals
Locations (1):
- Alfred Hospital, Melbourne, Australia